CLINICAL TRIAL: NCT02572063
Title: Omics4Aging: Stratification of Frailty Population Based on Nutrients Profiling and Metabolic Profiling at Baseline
Brief Title: Omics4Aging: Stratification of Frailty Population
Acronym: ProAge
Status: Terminated | Type: Observational
Why Stopped: Terminated, prior to its planned completion as anticipated by the protocol.
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 14.02.NIHS
Record Dates: First submitted 2015-05-04; First posted 2015-10-08 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-05

CONDITIONS: Malnutrition; Intellectual Frailty of Aging; Bone Fragility
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples and feces
Oversight: Data Monitoring Committee: No

SUMMARY:
The overall objective of the study is to stratify a frailty population based on nutrients profiling (amino acids, vitamins, minerals, fatty acids) and metabolic profiling (low molecular weight metabolites in urine and plasma) at baseline.

DETAILED DESCRIPTION:
This exploratory study will investigate ways to better characterize the frailty phenotype by a combination of i) geriatric assessment (here only: frailty criteria according to Fried), ii) clinical surrogate markers (including those of inflammation), iii) body composition, iv) nutritional profiling, v) metabolite profiling using a metabolomics approaches.

ELIGIBILITY:
Inclusion Criteria:

Unless otherwise specified, subjects who fulfill all of the following will be included:

1. Caucasian
2. Male or female between the ages of 65 and 79 years old
3. Three or more Fried Frailty Criteria (as diagnosed by investigator)
4. Informed consent obtained

Exclusion Criteria:

Any of the following criteria would render a subject ineligible for inclusion:

1. Dementia (previously diagnosed by general practitioner)
2. Hb1c (glycate Haemoglobin) >7.5% (>58 mmol/mol).
3. End stage disease (1 year after last chemotherapy treatment for cancer)
4. Drug abuse (alcohol - assessed by investigator)
5. Medications: no antibiotic treatment (for at least 4 weeks), immune suppressants, and or chronic use of corticosteroids
6. Currently participating or having participated in another clinical or nutritional intervention trial during the last 3 month
7. Chronic active inflammatory disease (e.g. rheumatoid arthritis, vasculitis, lupus erythematosus and Crohn's disease)
8. Chronic Active hepatitis
9. Kidney failure in Dialysis treatment
10. Any other condition that in the judgment of the lead investigator would not allow the subject to complete the study protocol

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 50 frail elderly free living healthy individuals, males and females, age 65-79.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-11-15 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
Comparison of Metabonomics, at baseline, among frail population. | 1 year
  Analysis of Metabolites in blood

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Capri, PhD, Principal Investigator — University of Bologna
Locations (1):
- Dr. Miriam Capri, Bologna, Italy